CLINICAL TRIAL: NCT01539772
Title: PITT0112: Becker Muscular Dystrophy - A Natural History Study to Predict Efficacy of Exon Skipping
Brief Title: Becker Muscular Dystrophy - A Natural History Study to Predict Efficacy of Exon Skipping
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Other Study IDs: PITT0112
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Becker Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Becker: BMD participants over 4 years of age with in-frame deletions in the dystrophin gene.
  .

SUMMARY:
This is a multi-center natural history study that will be conducted at participating centers in the Cooperative International Neuromuscular Research Group (CINRG). Following a baseline evaluation, participants will have three follow-up visits over a three-year period. The investigators will characterize the Becker muscular dystrophy phenotype, and correlate specific abnormal dystrophin proteins with the range of clinical outcomes.

DETAILED DESCRIPTION:
We will utilize the Cooperative International Neuromuscular Research group (CINRG) network to collect cohorts of Becker muscular dystrophy (BMD) patients with in-frame deletions in the dystrophin gene. We will collect clinical data across multiple body systems and correlate these findings to the high-resolution deletion break-point mapping performed from the tissue samples. We will investigate the observed variability to deepen our understanding of molecular mechanisms relevant to the optimization of exon skipping therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 4 or older
* Diagnosis of BMD with an in-frame deletion in the dystrophin gene, where the boundaries of the mutations are confirmed.

Exclusion Criteria:

• Investigator assessment of inability to comply with protocol

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BMD participants over 4 years of age with in-frame deletions in the dystrophin gene.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2012-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Strength and function | Annual
Quality of life | Annual
  These questionnaires include:
  * Pediatric Quality of Life Inventory (PedsQL)
  * Pediatrics and Adult Neuromuscular module Quality of Life (NeuroQOL)
Medical history assessment - ambulation status, medication history, hospitalizations, surgeries, nutrition, fractures, and cardiac tests | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Paula R Clemens, MD, Study Chair — University of Pittsburgh
Locations (16):
- United States (13):
  - University of California Davis, Sacramento, California
  - Children's National Health System, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- Alberta Children's Hospital, Calgary, Alberta, Canada
- Centro Clinico Nemo, Milan, Italy
- Institute of Genetic Medicine - Newcastle University, Newcastle upon Tyne, United Kingdom